CLINICAL TRIAL: NCT05627778
Title: A Head-to-head Comparison of 68Ga-P15-041 and 68Ga-PSMA-11 PET/CT Imaging in the Same Group of Prostate Bone Metastasis
Brief Title: 68Ga-P15-041 and 68Ga-PSMA-11 PET/CT Imaging in the Same Group of Prostate Bone Metastasis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-NM-11/041
Record Dates: First submitted 2022-11-08; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA-11 and 68Ga-P15-041 PET/ CT scan (Experimental): Patients of Prostate cancer PET/CT imaging: In two consecutive days each patient underwent a PET/ CT scan after intravenous administration of 68Ga- PSMA-11 and 68Ga-P15-041, respectively.
  Interventions: Drug: 68Ga-PSMA-11; Drug: 68Ga-P15-041

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — Intravenous injection of one dosage of 148-185 MBq (4-5 mCi) 68Ga-PSMA-11. Tracer doses of 68Ga- PSMA-11 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: 68Ga-PSMA-11 injection
Drug: 68Ga-P15-041 — Intravenous injection of one dosage of 148-185 MBq (4-5 mCi) 68Ga-P15-041. Tracer doses of 68Ga- 15-041 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: 68Ga-P15-041 injection

SUMMARY:
Tumor bone metastasis refers to the metastasis of malignant tumors to the bone through lymph, blood or direct invasion to generate daughter tumors, which is the most common bone tumor. More than 40% of patients with malignant tumors will have bone metastasis, among which breast cancer, prostate cancer is more common, once the tumor cells occur bone metastasis, it means that the disease enters the advanced stage, posing a serious threat to the life safety of patients, therefore, early diagnosis of various primary malignant tumor bone metastases, can lay the foundation for clinical implementation of effective treatment measures. The laboratory of Hank F. Kung at the University of Pennsylvania has developed a new generation of 68Ga-labeled radiopharmaceutical P15-041 ([68Ga]Ga-HBED-CC-BP) based on existing phosphonate-targeting molecular probes (Figure 1). Data from preclinical studies indicate that P15-041 shows additional advantages in rapid and easy complex formation compared to current [68Ga]Ga-BPAMD, [68Ga]Ga-NO2AP-BP, [68Ga]Ga-DOTA- (ZOL). In vivo experiments, P15-041 showed good bone resorption and rapid renal excretion in normal mice. Haiyan Hong et al. [13] prepared multiple clinical doses of P15-041 and successfully evaluated it in patients, followed by intravenous P15-041, followed by a whole body PET/CT scan. Robert K. Doot et al. conducted dosimetric experiments on P15-041, analyzed the radioactive distribution of the drug in normal organs and the dynamic change of the dose of the drug in the body over time, and the results showed that P15-041 had high uptake in the bladder wall and bone cortex, blood and other tissues cleared quickly, and there was obvious radioactive enrichment in the myocardium in the early stage of imaging, and P15-041 had the potential to become a new generation of excellent phosphonate molecular probes.

DETAILED DESCRIPTION:
Tumor bone metastasis (Tumor Bone Metastasis) refers to the metastasis of malignant tumor to the bone through lymphatic, blood or direct infiltration, resulting in sub-tumor, which is the most common bone tumor. More than 40% of patients with malignant tumors will develop bone metastasis, among which breast cancer and prostate cancer are more common. Once bone metastasis occurs in tumor cells, it means that the disease has entered an advanced stage and poses a serious threat to the life safety of patients. Therefore, early diagnosis Bone metastases from various primary malignant tumors can lay the foundation for the clinical implementation of effective treatment measures. At present, single photon emission computer-aided tomography (SPECT) technetium-99 (99mTc)-methylenediphos-phonate (MDP) is the preferred method for early diagnosis of tumor bone metastases , but benign bone Disease (such as bone degeneration, trauma, inflammatory response) and reactive changes during treatment ((scintillation phenomenon) can also be manifested as abnormal radioactive concentrations, with the possibility of false positives . Positron emission tomography Imaging (PET) technology is a nuclear medicine imaging method that integrates anatomical images of diseases and functional metabolism. It combines radioisotopes with compounds to achieve the function of imaging the metabolism of targeted substances. Compared with other imaging methods, PET molecular probes have higher sensitivity. Clinically, [18F]F-FDG PET/CT is commonly used to observe the metabolic status of bone metastases, which can show bone metastases that have not yet undergone osteogenesis or osteolysis. Vine-labeled phosphonates are bone imaging agents commonly used clinically to evaluate bone diseases such as infection (osteomyelitis), noninfectious inflammation (arthritis), trauma, metabolic bone disease, benign and malignant tumors, and metastases. ), the imaging agent reaches the bones of the whole body with the blood flow through intravenous injection, and is distributed in the bone tissue through ion exchange and chemical adsorption with the hydroxyapatite crystals in the bone, and the newly formed collagen has a higher effect on the bone imaging agent. Recent studies have shown that, the uptake mechanism of radionuclide-labeled phosphonates such as [99mTc]Tc-DPD, [99mTc]Tc-HMDP and [99mTc]Tc-PYP in amyloid myocardial deposition It is not fully understood, but some investigators have evaluated biopsies and found that microcalcifications are often present in cardiac amyloid deposits and may be associated with positive phosphonate imaging. However, [99mTc]Tc imaging agents are still not effective for Quantitative assessment of amyloid deposition. Recently, with the successful application of 68Ga-somatostatin receptor imaging agents in PET/CT, people have gradually shifted their attention to the "new generation" positron nuclides 68Ga, 68Ge /68Ga radionuclide generator can prepare 68Ga based PET tracer without adjacent cyclotron, in addition, 68Ga excellent physical properties (t1/2: 68min; 89%β+, 1.92mev maximum energy) Suitable for PET imaging, therefore, the development of bisphosphonates labeled with 68Ga will meet the need for a source of PET tracers.

Based on the existing phosphonate-targeted molecular probes, the Hank F. Kung laboratory at the University of Pennsylvania has developed a new generation of 68Ga-labeled radiopharmaceutical P15-041 ([68Ga]Ga-HBED-CC-BP). Preclinical data show that P15-041 exhibits rapid and facile complex formation compared to current [68Ga]Ga-BPAMD, [68Ga]Ga-NO2AP-BP, [68Ga]Ga-DOTA-(ZOL) an additional advantage. In in vivo experiments, P15-041 exhibited good bone resorption and rapid renal excretion in normal mice. Haiyan Hong et al. [13] prepared various clinical doses of P15-041 and successfully evaluated them in patients who performed whole-body PET/CT scans after intravenous administration of P15-041. Robert K. Doot et al conducted a dosimetry test on P15-041, and analyzed the radioactive distribution of the drug in normal organs and the dynamic changes of the drug in vivo with time. The cortical bone uptake is high, the blood and other tissues are cleared quickly, and there is obvious radioactive enrichment in the myocardium in the early stage of imaging. P15-041 has the potential to become a new generation of excellent phosphonate molecular probes.

ELIGIBILITY:
Inclusion Criteria:

* confirmed suspected prostate bone metastasis patients;
* 68Ga-PSMA-11 and 68Ga-P15-041 PET/CT within one week;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
detection capability of bone metastasis | through study completion, an average of 1 year
  the bone metastasis number detected by 68Ga-P15-041 PET/CT for prostate cancer in comparison with 68Ga-PSMA-11 PET/ CT
SUVmax of bone metastasis | through study completion, an average of 1 year
  the tumor uptake on 68Ga-P15-041 PET/CT for prostate cancer in comparison with 68Ga-PSMA-11 PET/CT

SECONDARY OUTCOMES:
PSMA expression and SUV | through study completion, an average of 1 year
  Correlation between PSMA expression and SUV in PET

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Doc., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China